CLINICAL TRIAL: NCT05667753
Title: Large-scale Implementation of a mHealth Obesity Prevention Program Within Swedish Primary Child Healthcare: MINISTOP 3.0 Study Protocol
Brief Title: Large Scale Implementation of MINISTOP 3.0
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Christine Delisle Nyström, Docent, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-01710-01
Record Dates: First submitted 2022-12-19; First posted 2022-12-29 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Obesity, Child
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial utilizing a hybrid type III implementation-effectiveness design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Basic (Active Comparator): The MINISTOP app will be offered to all parents of children at the 2.5/3-year routine visit at primary child healthcare. The child healthcare centers randomly allocated to the basic group will receive the basic implementation strategy package.
  Interventions: Behavioral: MINISTOP 3.0
- Enhanced (Experimental): The MINISTOP app will be offered to all parents of children at the 2.5/3-year routine visit at primary child healthcare. The child healthcare centers randomly allocated to the enhanced group will receive the enhanced implementation strategy package.
  Interventions: Behavioral: MINISTOP 3.0

INTERVENTIONS:
Behavioral: MINISTOP 3.0 — MINISTOP 3.0 is a behavioral changed program with the overall aim to promote healthier lifestyle behaviors (i.e., diet, physical activity, and sedentary behavior) among 2.5/3-year old children. The MINISTOP 3.0 program consists of features such as information, monitoring, and feedback (dietary variables, physical activity, and screen time) and is built around 13 themes over a 6-month period.

SUMMARY:
MINISTOP is an evidence-based app for parents of preschool aged children with the overall aim to promote healthy lifestyle behaviors and prevent the development of overweight and obesity. MINISTOP has been previously been evaluated in two previous trials (MINISTOP 1.0 and 2.0) with promising results. Therefore, the overall aim of this trial is to evaluate the large scale implementation of MINISTOP within Swedish primary child healthcare. The specific aims are to:

(i) To compare two different implementation strategies for MINISTOP 3.0 (i.e., Basic vs.

Enhanced) on: a) acceptability, appropriateness, feasibility as well as organizational readiness to implement MINISTOP 3.0 within primary child healthcare (primary outcomes) and b) reach, costs, adoption, and sustainability of MINISTOP 3.0 within primary child healthcare (secondary outcomes).

(ii) To compare two different implementation strategies of MINISTOP 3.0 within primary child healthcare on children's key dietary indicators, physical activity, and screen time (secondary outcomes).

(iii) To compare the cost-effectiveness of two different implementation strategies for MINISTOP 3.0.

ELIGIBILITY:
Inclusion Criteria:

* Child healthcare nurse at participating child healthcare centers

No exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in acceptability of MINISTOP 3.0 | Baseline, 3 &12 months after implementation
  Acceptability of MINISTOP 3.0 by child healthcare nurses (assessed by the questionnaire by Weiner et al.). It includes four questions assessed on a five point likert scale ranging from completely disagree to completely agree.
Change in appropriateness of MINISTOP 3.0 | Baseline, 3 & 12 months after implementation
  Appropriateness of MINISTOP 3.0 by child healthcare nurses (assessed by the questionnaire by Weiner et al.). It includes four questions assessed on a five point likert scale ranging from completely disagree to completely agree.
Change in feasibility of MINISTOP 3.0 | Baseline, 3 &12 months after implementation
  Feasibility of MINISTOP 3.0 by child healthcare nurses (assessed by the questionnaire by Weiner et al.). It includes four questions assessed on a five point likert scale ranging from completely disagree to completely agree.
Change in organizational readiness for implementing MINISTOP 3.0 | Baseline 3 and 12 months after implementation
  Organizational readiness as perceived by child healthcare nurses, which will be measured using the E-READY questionnaire. This questionnaire consists of 32 questions rated on a 4-point likert scale.

SECONDARY OUTCOMES:
Adoption of MINISTOP 3.0 | 3, 8, and 12 months after implementation
  Assessment based on a questionnaire from 1 to 5 with 5 indicating a better score
Costs of the implementation of MINISTOP 3.0 | Baseline and 2, 4, 6, 8, 10, and 12 months after implementation.
  Collected through administrative data from participating child healthcare centers regarding implementing and maintaining the MINISTOP platform, as well as the nurses time with the MINISTOP program (Swedish Krona, SEK).
Sustainability | 12 months after implementation
  Semi-structured interviews with primary child healthcare nurses
Parental usage of MINISTOP 3.0 using objectively measured activity in the app | 6 months after the families start using the MINISTOP app
  Number of recordings and messages read in the app (per time unity such as per week)
Children's intake of key dietary indicators as assess by a questionnaire. | Baseline and 6 months after receiving MINISTOP 3.0
  Intake of fruits, vegetables, sweet and savoury snacks, as well as sweetened beverages (grams/day)
Children's physical activity as assessed by a questionnaire | Baseline and 6 months after receiving MINISTOP 3.0
  Time spent in moderate-to-vigorous physical activity (minutes/day)
Children's screen time as assessed by a questionnaire | Baseline and 6 months after receiving MINISTOP 3.0
  Time spent watching screens (minutes/day)

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Huddinge, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thomas K, Lof M, Lundgren M, Fagerstrom M, Hesketh KD, Brown V, Habel H, Delisle Nystrom C. MINISTOP 3.0: Implementation of a mHealth obesity prevention program within Swedish child healthcare - study protocol for a cluster randomized controlled trial. BMC Public Health. 2024 Sep 27;24(1):2594. doi: 10.1186/s12889-024-20137-0. PMID 39333981